CLINICAL TRIAL: NCT03344731
Title: Cognitive Abilities in Brain Damaged Patients
Acronym: Cog
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Neuromed IRCCS (Other)
Responsible Party: Principal Investigator, Mario Stampanoni Bassi, Principal Investigator, Neuromed IRCCS
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Basic Science
Other Study IDs: Neuromed_Cog
Record Dates: First submitted 2017-10-20; First posted 2017-11-17 (Actual); Last update posted 2022-10-31 (Actual); Status verified 2022-10

CONDITIONS: Brain Damage
MeSH Terms: conditions — Brain Injuries

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental Group (Experimental): Patient with any form ob brain damage
  Interventions: Behavioral: Cognitive evaluation; Device: Non-invasive brain stimulation
- Control Group (Other): Healthy volounteers
  Interventions: Behavioral: Cognitive evaluation; Device: Non-invasive brain stimulation

INTERVENTIONS:
Behavioral: Cognitive evaluation — Cognitive task
Device: Non-invasive brain stimulation — Transcranial Magnetic Stimulation (TMS)

SUMMARY:
The presence of damage to the central and / or peripheral nervous system resulting from pathologies of a different nature (such as multiple sclerosis, Parkinson's disease, dementia, cranial trauma, stroke, epilepsy or other neurological syndromes) is commonly a cause of physical and mental disability. The presence of memory or language cognitive deficits is often evident at a first clinical examination. However, difficulties in cognitive areas such as decision-making, social and emotional cognition or particular forms of learning may be less evident, while exerting a strong impact on the quality of life of patients.

The main purpose of this proposal is to investigate cognitive abilities in patients with neurological damage, through a series of specific tasks.

In addition, the contribution of specific brain areas to the cognitive tasks will be assessed by direct modulation of brain activity. This modulation will be achieved by using non-invasive brain stimulation techniques such as Transcranial Magnetic Stimulation (TMS) and Direct Transcranial Electric Stimulation (tDCS).

DETAILED DESCRIPTION:
The presence of damage to the central and / or peripheral nervous system resulting from pathologies of a different nature (such as multiple sclerosis, Parkinson's disease, dementia, cranial trauma, stroke, epilepsy or other neurological syndromes) is commonly a cause of physical and mental disability. The presence of memory or language cognitive deficits is often evident at a first clinical examination. However, difficulties in cognitive areas such as decision-making, social and emotional cognition or particular forms of learning may be less evident, while exerting a strong impact on the quality of life of patients.

The main purpose of this proposal is to investigate cognitive abilities in patients with neurological damage, through a series of specific tasks. To this end, a series of tests and questionnaires will be used, described in detail below, to evaluate various cognitive functions, including decision-making, problem-solving, learning, memory, executive, social and emotional cognition.

In addition, the contribution of specific brain areas to the cognitive tasks will be assessed by direct modulation of brain activity. This modulation will be achieved by using non-invasive brain stimulation techniques such as Transcranial Magnetic Stimulation (TMS) and Direct Transcranial Electric Stimulation (tDCS).

TMS, in particular, is a non-invasive neuronal stimulation of surface areas of the brain that since its inception has been frequently used in neurology as a diagnostic and research tool. TMS uses magnetic fields to induce electrical currents that facilitate or inhibit cortical activity. TDCS consists in the application of weak electrical currents to generate an electric field that can modulate neural activity in an excitatory or inhibitory manner. TMS and tDCS can be used in the experimental field to modulate cortical activity and modify performance during cognitive tasks.

An important mechanism responsible for clinical, cognitive and functional recovery after neurological damage of different types is synaptic plasticity. Nervous tissue has the ability to permanently enhance or de-energize inter-neuronal transmission at synaptic level. By increasing the efficiency of synaptic transmission, through a phenomenon known as long-term potentiation (LTP), it is possible to compensate the loss of synaptic pulses on survived neurons due to brain damage and restore their function. LTP is also capable of guiding the formation of new brain circuits (structural plasticity), with compensatory and adaptive function . Indeed, neurotransmitters, in addition to their bioelectric conduction activity, also act on neurotrophic factors.

Aim The aim of this study is to evaluate cognitive abilities in healthy subjects and in patients with neurological injury of various kinds (such as multiple sclerosis, Parkinson's disease, dementia, cranial trauma, stroke, epilepsy or other neurological syndromes) as well as to deepen the contribution of specific brain areas in carrying out these cognitive tasks. This will be made possible thanks to the specific skills of a multidisciplinary team of neurologists and physiatrists, health professionals such as physiotherapists, occupational therapists, psychologists, speech therapists, and the support of a biomedical engineer. These professional figures are already available at the UUOOCC of Neurology Neurosurgery and Neurosurgery directed by the proposer.

ELIGIBILITY:
Inclusion criteria:

* Males or females aged between 18 and 80;
* Presence of brain damage resulting from: Multiple Sclerosis, Parkinson Disease, Dementia, Cranial Trauma, Neurosurgical Intervention, Ictus, Epilepsy or Other Neurological Syndromes (for the experimental group only);
* Absence of neurological disorders (for the control group only);
* be able to follow the protocol's directions throughout the study;
* Female subjects undertake not to schedule a pregnancy for the duration of the study;
* Patients should be able to follow protocol guidelines throughout the study;
* Patients should be able to understand the aims and risks of the study;
* Signature of informed consent, approved by our Ethics Committee.

Exclusion criteria:

* Incapability even partial to understand and want;
* Patients with other pathologies which, according to the opinion of the scientific manager, prevent the recruitment;
* When using non-invasive brain stimulation techniques or subjects should not submit any of their own contraindications (for further details, see the "Methods" and "Stimulation Evaluation Questionnaire" attached to this proposal);
* Pregnancy, breastfeeding, and delivery not less than three months before the start of the study.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2017-12-15 (Actual); Primary Completion 2024-12-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Learning | up to 3 years
  Associative learning tasks will be inspired by those previously used in literature during which subjects should learn a series of stimulus-outcome associations (pavlovian learning) or response-outcome (instrumental learning).
Risk decision-making | up to 3 years
  Neurological deficits can affect the ability to learn from past mistakes and make decisions for the future. To observe the decision-making mechanisms and to analyze the ability to choose, a series of more or less risky economic choices will be presented, which can result in both a payout or a loss. Initially participants receive a sum of virtual money with the instruction to maximize the payout. An unaltered decision skill should have the ability to make the least risky choice and involve more long-term wins.
Social and emotional cognition | up to 3 years
  To evaluate social and emotional cognition, a series of tests will be used to quantify both the ability to empathize and understand the emotions of others, and the ability to intrepret their thoughts and intentions. A classical test involves the presentation of facial expressions and is asked to choose which word best describes what the person in the image is thinking or trying.

CONTACTS AND LOCATIONS:
Overall Officials: Diego Centonze, MD, Principal Investigator — IRCCS Neuromed
Locations (1):
- IRCCS Neuromed, Pozzilli, Isernia, Italy

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Chen R, Classen J, Gerloff C, Celnik P, Wassermann EM, Hallett M, Cohen LG. Depression of motor cortex excitability by low-frequency transcranial magnetic stimulation. Neurology. 1997 May;48(5):1398-403. doi: 10.1212/wnl.48.5.1398. PMID 9153480
- [Result] Chiaravalloti ND, DeLuca J. Cognitive impairment in multiple sclerosis. Lancet Neurol. 2008 Dec;7(12):1139-51. doi: 10.1016/S1474-4422(08)70259-X. PMID 19007738
- [Result] Fortin S, Godbout L, Braun CM. Cognitive structure of executive deficits in frontally lesioned head trauma patients performing activities of daily living. Cortex. 2003 Apr;39(2):273-91. doi: 10.1016/s0010-9452(08)70109-6. PMID 12784889
- [Result] Jochumsen M, Signal N, Nedergaard RW, Taylor D, Haavik H, Niazi IK. Induction of Long-term Depression-like Plasticity by Pairings of Motor Imagination and Peripheral Electrical Stimulation. Front Hum Neurosci. 2015 Dec 1;9:644. doi: 10.3389/fnhum.2015.00644. eCollection 2015. PMID 26648859
- [Result] Rossini PM, Burke D, Chen R, Cohen LG, Daskalakis Z, Di Iorio R, Di Lazzaro V, Ferreri F, Fitzgerald PB, George MS, Hallett M, Lefaucheur JP, Langguth B, Matsumoto H, Miniussi C, Nitsche MA, Pascual-Leone A, Paulus W, Rossi S, Rothwell JC, Siebner HR, Ugawa Y, Walsh V, Ziemann U. Non-invasive electrical and magnetic stimulation of the brain, spinal cord, roots and peripheral nerves: Basic principles and procedures for routine clinical and research application. An updated report from an I.F.C.N. Committee. Clin Neurophysiol. 2015 Jun;126(6):1071-1107. doi: 10.1016/j.clinph.2015.02.001. Epub 2015 Feb 10. PMID 25797650
- [Result] Schrag A, Jahanshahi M, Quinn N. What contributes to quality of life in patients with Parkinson's disease? J Neurol Neurosurg Psychiatry. 2000 Sep;69(3):308-12. doi: 10.1136/jnnp.69.3.308. PMID 10945804